CLINICAL TRIAL: NCT06751251
Title: The Exploration of OX40 (CD134) Expression Levels in Sarcoma Specimens and Its Clinical Application in Prognosis Determination
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Principal Investigator, Peking University People's Hospital
Other Study IDs: PKUPH-sarcoma 20
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Biomarkers; Progression
Keywords: Sarcoma; OX40; Transcriptomics; Biomarker; CD134; prognosis
MeSH Terms: conditions — Sarcoma; Disease Progression | interventions — RNA-Seq

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OX40 (CD134) expression levels of sarcoma specimens in treatment-native sarcoma patients: Before delivering neoadjuvant chemotherapy, using IHC to test the protein expression of OX40 and using RNA-seq to test the RNA of OX40
  Interventions: Diagnostic Test: IHC: Immunohistochemistry; Genetic: RNA-seq
- OX40 (CD134) expression levels of sarcoma specimens in chemotherapy treated sarcoma patients: After neoadiuyant chemotherapy, using IHC to test the protein expression of OX40 and using RNA-seq to test the RNA of OX40
  Interventions: Diagnostic Test: IHC: Immunohistochemistry; Genetic: RNA-seq

INTERVENTIONS:
Diagnostic Test: IHC: Immunohistochemistry — Immunohistochemistry will be implied in tissue sections to test the expression of OX4O in sarcoma.
Genetic: RNA-seq — RNA-seq will be implied in tissue sections to test the expression of CD134 RNA expression in sarcoma.

SUMMARY:
This study aims to investigate the expression of OX40 (CD134) in sarcomas and its impact on prognosis, with the goal of identifying novel biomarkers for early resistance detection and optimizing treatment strategies for sarcoma patients. Sarcomas are a highly heterogeneous group of malignant tumors, for which current treatment options are often suboptimal in certain patients, and effective biomarkers to guide therapy are lacking. As a T-cell costimulatory receptor, OX40 plays a significant role in immune regulation across various solid tumors and holds promise as a potential therapeutic target.

The researcher's team has previously identified high OX40 expression in sarcomas through database analysis and validated the therapeutic efficacy of antibody-drug conjugates targeting OX40 in in vivo experiments using sarcoma cell lines in murine models. This study will evaluate the mRNA expression levels of OX40 in tumor tissues from sarcoma patients and assess OX40 protein expression using immunohistochemical staining. By integrating these findings with clinical and pathological data, the study will explore the potential of OX40 expression levels in tumor tissues as biomarkers for predicting treatment response and prognosis in primary bone tumors. The results aim to provide scientific evidence for the clinical application of OX40-targeted therapies and to propose novel therapeutic strategies to improve survival outcomes in sarcoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8 years or older.
* Diagnosed with high-grade osteosarcoma or Ewing sarcoma, confirmed through clinical evaluation or histopathological examination. For patients with localized tumors or solitary pulmonary lesions, pathological confirmation is required; for patients with multiple pulmonary metastases, pathological examination is not necessary.
* Treatment-naïve patients who have not received standard first-line chemotherapy regimens for osteosarcoma or Ewing sarcoma.(First-line chemotherapy drugs include high-dose methotrexate, anthracyclines, cisplatin, and ifosfamide. For Ewing sarcoma, the standard first-line regimen is VDC followed by IE.)
* All other examination indicators suggest that the patient is eligible for standardized chemotherapy and surgical treatment for bone tumors.

Exclusion Criteria:

* Inability to undergo standardized chemotherapy and surgical treatment for bone tumors at this center.
* Refusal to adhere to follow-up according to standardized diagnostic and treatment protocols.
* Any condition that, in the investigator's opinion, may harm the participant or prevent them from meeting or complying with the study requirements.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initial treated osteosarcoma patients in PKUPH and later would recieve definitive surgery in PKUPH with complete clinical materials.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
correlation of quantity of Protein OX40 Expression with clinical evaluation | 6 months
  Clinical evaluation according to RECIST 1.1

SECONDARY OUTCOMES:
correlation of quantity of CD134 RNA with event-free survival | 6 months
  correlation of quantity of CD134 RNA with event-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thapa B, Kato S, Nishizaki D, Miyashita H, Lee S, Nesline MK, Previs RA, Conroy JM, DePietro P, Pabla S, Kurzrock R. OX40/OX40 ligand and its role in precision immune oncology. Cancer Metastasis Rev. 2024 Sep;43(3):1001-1013. doi: 10.1007/s10555-024-10184-9. Epub 2024 Mar 25. PMID 38526805
- [Background] Xie L, Guo W, Wang Y, Yan T, Ji T, Xu J. Apatinib for advanced sarcoma: results from multiple institutions' off-label use in China. BMC Cancer. 2018 Apr 6;18(1):396. doi: 10.1186/s12885-018-4303-z. PMID 29625604